CLINICAL TRIAL: NCT04814862
Title: Descriptive and Risk Factor Analysis of Neuropsychiatric and Neurodevelopmental Disorders in Children With Systemic Inflammatory Disease
Brief Title: Neurodevelopmental Disorders in Children With Systemic Inflammatory Disease
Acronym: Artemis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210146; IDRCB: 2020-A02841-38 (Other: ANSM)
Record Dates: First submitted 2021-03-19; First posted 2021-03-24 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-03

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Spermine Synthase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: 3 validated questionnaires (ADHD-RS, SRS, BRIEF) for the diagnosis of neurodevelopmental disorders — Completion of three validated questionnaires for the diagnosis of neurodevelopmental disorders

SUMMARY:
Systemic inflammatory diseases in children include autoinflammatory diseases (deregulation of the innate immune system with production of pro-inflammatory cytokines) and autoimmune diseases (deregulation of the adaptive immune system with production of pathogenic autoantibodies). Neurological damage has been reported in both cases, but the neurodevelopmental psychiatric manifestations are poorly known, especially in children.

Neurodevelopmental disorders are a broad spectrum of pathologies that are underpinned by common symptomatic dimensions. They have a common physiopathology combining genetic predisposing factors as well as environmental risk factors, making it possible to study them from a global point of view. Among the environmental risk factors, the immune system seems to play an important role in the appearance of these pathologies.

In recent years, fundamental and animal studies have pointed to an important role of the immune system at the cerebral level. Indeed, far from the old notion of ""immune privilege"", the innate or adaptive immune balance seems to have a fundamental role in the proper development and functioning of the brain. Consequently, any modification of the immune balance could then disrupt neurodevelopment. Indeed, in recent years epidemiological studies seem to indicate the role of immune-mediated events during pregnancy (maternal autoimmune/inflammatory pathology or infection during pregnancy) or the first years of life (autoimmune/inflammatory pathology) as risk factors for neurodevelopmental disorders. Neurodevelopmental manifestations are very poorly known in systemic inflammatory pathologies. They can have a significant impact and justify adapted care in order to limit the functional impact. The main objective of our study will be to define the prevalence of neurodevelopmental disorders in children with systemic inflammatory diseases.

DETAILED DESCRIPTION:
Systemic inflammatory diseases in children include auto-inflammatory diseases (deregulation of the innate immune system with production of pro-inflammatory cytokines) and autoimmune diseases (deregulation of the adaptive immune system with production of pathogenic autoantibodies). Neurological damage has been reported in both cases, but the neurodevelopmental psychiatric manifestations are poorly known, especially in children. Neurodevelopmental disorders are a broad spectrum of pathologies with common symptomatic dimensions. They present a common physiopathology combining genetic predisposition factors as well as environmental risk factors, which allows them to be studied from a global perspective. Among the environmental risk factors, the immune system seems to play an important role in the appearance of these pathologies. In recent years, fundamental and animal studies have highlighted an important role of the immune system at the cerebral level. Indeed, far from the old notion of ""immune privilege"", the innate or adaptive immune balance seems to have a fundamental role in the proper development and functioning of the brain. Consequently, any change in the immune balance could then disrupt neurological development. Indeed, in recent years, epidemiological studies seem to indicate the role of immune-mediated events during pregnancy (maternal autoimmune/inflammatory pathology or infection during pregnancy) or the early years of life (autoimmune/inflammatory pathology) as risk factors for neurodevelopmental disorders.

Neurodevelopmental manifestations are very poorly known in systemic inflammatory pathologies. They can have a significant impact and justify adapted care in order to limit the functional impact. Indeed, due to their pathology, these patients produce pro-inflammatory cytokines at an early stage which could have an impact on their neurodevelopment. The identification of neurodevelopmental disorders in these patients could be a clinical and epidemiological validation of preclinical studies highlighting the importance of the immune system in the proper development of the brain. The main objective of our study will be to define the prevalence of neurodevelopmental disorders in children suffering from systemic inflammatory diseases via the passing on by parents of children between 5 and 17 years old of three hetero-questionnaires (i) SRS (assessing social interaction disorders), (ii) ADHD-RS (assessing attentional and hyperactivity difficulties) (iii) BRIEF (assessing difficulties in executive functions). All the results of these scales are adjusted for the age and sex of the patients and provide a T-score (allowing a valid comparison).

This is a multi-centre cross-sectional study involving the collection of data from patients' medical records and questionnaires from patients' parents.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a systemic inflammatory disease
* Age between 5 and 17 years old
* Parents informed and having signed a consent or having consented orally in case of absence of one of the two parents

Exclusion Criteria:

* Insufficient comprehension of the French language
* Mental retardation with IQ <30
* Not affiliated to a social security system

Ages: 5 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: All pediatric patients with systemic inflammatory disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-12-06 (Estimated); Primary Completion 2022-12-06 (Estimated); Study Completion 2022-12-06 (Estimated)

PRIMARY OUTCOMES:
To define the prevalence of neurodevelopmental disorders in children with systemic inflammatory disease. | 1 day
  Number of children scoring above 75th percentile on ADHD-RS out of all patients presenting a systemic inflammatory pathology.
  All the results of these scales are adjusted for the age and sex of the patients (allowing a valid comparison).

SECONDARY OUTCOMES:
To define the prevalence of neurodevelopmental disorders in children with systemic inflammatory disease. | 1 day
  Number of children scoring T-score above 60 on SRS out of all patients presenting a systemic inflammatory pathology.
  All the results of this scale are adjusted for the age and sex of the patients (allowing a valid comparison).
To define the prevalence of neurodevelopmental disorders in children with systemic inflammatory disease. | 1 day
  Number of children scoring above 1SD on BRIEF out of all patients presenting a systemic inflammatory pathology.
  All the results of this scale are adjusted for the age and sex of the patients (allowing a valid comparison).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MELKI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No